CLINICAL TRIAL: NCT00775749
Title: Transdermal Nicotine in Female Patients at High Risk for PONV
Brief Title: Transdermal Nicotine in Female Patients at High Risk for Post Operative Nausea and/or Vomiting (PONV)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study is not feasible with the number of subjects needed to complete it.
Sponsor: Ochsner Health System (Other)
Responsible Party: Principal Investigator, Stuart Hart, Director of Obstetric Anesthesiology, Ochsner Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PONV
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Postoperative Nausea and Vomiting
Keywords: post operative nausea and vomiting; gynecological surgery; outpatient surgery; nicotine patch; laparoscopic surgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Vomiting | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The nicotine patch will be applied prior to surgery and remain on the right upper back for 24 hours.
  Interventions: Drug: transdermal nicotine patch
- 2 (Placebo Comparator): The placebo patch has no active ingredients and the same inactive ingredients as the nicotine patch. It will be administered the same fashion as the nicotine patch.
  Interventions: Drug: placebo patch

INTERVENTIONS:
Drug: transdermal nicotine patch — The 7 mg transdermal nicotine patch will be applied to the right upper back prior to surgery. It will be covered with an opaque bandage to minimize inadvertent removal and conceal which patch has been placed.
  Other Names: Nicoderm CQ Step 3
  Arms: 1
Drug: placebo patch — The placebo patch will be applied to the right upper back prior to surgery. It will be covered with an opaque bandage to minimize inadvertent removal and conceal which patch has been placed.
  Other Names: Tegaderm patch
  Arms: 2

SUMMARY:
The purpose of this study is to see if the nicotine patch reduces post operative nausea and/or vomiting (PONV) among non-smoking patients who are at high risk of PONV.

DETAILED DESCRIPTION:
There are certain known risk factors for post-operative nausea and/or vomiting: the use of opioids during surgery, female gender, laparoscopic surgery, gynecologic surgery, strabismus repair, the use of a general anesthetic, obesity, and non-smoker. Patients with four or more of these risk factors have an 80% occurrence rate of post-operative nausea and/or vomiting and are classified as "high risk". It has been shown that those who use tobacco have about a 50% reduction in post-operative nausea and/or vomiting.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* female
* health patient or acute illness
* undergoing outpatient-type general surgery, especially those associated with increased incidence of post-operative nausea and/or vomiting such as gynecological procedures
* undergoing general anesthesia for the surgery
* receiving opioids during surgery
* non-smokers

Exclusion Criteria:

* history of any heart condition
* history of uncontrolled hypertension, or presence of any condition that could be made drastically worse by an increase in blood pressure
* history of an aneurysm
* active tobacco use within the past five years
* works or lives in the presence of cigarette smoke
* pregnant
* mentally ill
* prisoners
* history of allergic reaction to nicotine or to adhesive patches
* history of allergic reaction to propofol, versed, fentanyl, zofran, decadron, and reglan

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is whether the patient experienced post-operative nausea and/or vomiting. | The outcome measure will be assessed within 24 hours after the application of the patch.

SECONDARY OUTCOMES:
The secondary outcome is to assess how many episodes of post-operative nausea and/or vomiting the patient experiences. | The outcome measure will be assessed within 24 hours of the application of the patch.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart R Hart, M.D., Principal Investigator — Ochsner Health Systems; Heather S Porter, Study Director — Ochsner Health Systems
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Joseph AM, Fu SS. Safety issues in pharmacotherapy for smoking in patients with cardiovascular disease. Prog Cardiovasc Dis. 2003 May-Jun;45(6):429-41. doi: 10.1053/pcad.2003.YPCAD14. PMID 12800126
- [Background] Joseph AM, Norman SM, Ferry LH, Prochazka AV, Westman EC, Steele BG, Sherman SE, Cleveland M, Antonuccio DO, Hartman N, McGovern PG. The safety of transdermal nicotine as an aid to smoking cessation in patients with cardiac disease. N Engl J Med. 1996 Dec 12;335(24):1792-8. doi: 10.1056/NEJM199612123352402. PMID 8943160
- [Background] Tzivoni D, Keren A, Meyler S, Khoury Z, Lerer T, Brunel P. Cardiovascular safety of transdermal nicotine patches in patients with coronary artery disease who try to quit smoking. Cardiovasc Drugs Ther. 1998 Jul;12(3):239-44. doi: 10.1023/a:1007757530765. PMID 9784902
- [Result] Davidson M, Epstein M, Burt R, Schaefer C, Whitworth G, McDonald A. Efficacy and safety of an over-the-counter transdermal nicotine patch as an aid for smoking cessation. Arch Fam Med. 1998 Nov-Dec;7(6):569-74. doi: 10.1001/archfami.7.6.569. PMID 9821833
- [Result] Head KA, Jurenka JS. Inflammatory bowel disease Part 1: ulcerative colitis--pathophysiology and conventional and alternative treatment options. Altern Med Rev. 2003 Aug;8(3):247-83. PMID 12946238
- [Result] Flood P, Daniel D. Intranasal nicotine for postoperative pain treatment. Anesthesiology. 2004 Dec;101(6):1417-21. doi: 10.1097/00000542-200412000-00023. PMID 15564950
- [Result] Khoury Z, Comans P, Keren A, Lerer T, Gavish A, Tzivoni D. Effects of transdermal nicotine patches on ambulatory ECG monitoring findings: a double-blind study in healthy smokers. Cardiovasc Drugs Ther. 1996 May;10(2):179-84. doi: 10.1007/BF00823596. PMID 8842510
- [Result] Mahmarian JJ, Moye LA, Nasser GA, Nagueh SF, Bloom MF, Benowitz NL, Verani MS, Byrd WG, Pratt CM. Nicotine patch therapy in smoking cessation reduces the extent of exercise-induced myocardial ischemia. J Am Coll Cardiol. 1997 Jul;30(1):125-30. doi: 10.1016/s0735-1097(97)00128-9. PMID 9207632
- [Result] Richardson CE, Morgan JM, Jasani B, Green JT, Rhodes J, Williams GT, Lindstrom J, Wonnacott S, Peel S, Thomas GA. Effect of smoking and transdermal nicotine on colonic nicotinic acetylcholine receptors in ulcerative colitis. QJM. 2003 Jan;96(1):57-65. doi: 10.1093/qjmed/hcg007. PMID 12509650
- [Result] Shytle RD, Silver AA, Wilkinson BJ, Sanberg PR. A pilot controlled trial of transdermal nicotine in the treatment of attention deficit hyperactivity disorder. World J Biol Psychiatry. 2002 Jul;3(3):150-5. doi: 10.3109/15622970209150616. PMID 12478880
- [Result] Silver AA, Shytle RD, Philipp MK, Wilkinson BJ, McConville B, Sanberg PR. Transdermal nicotine and haloperidol in Tourette's disorder: a double-blind placebo-controlled study. J Clin Psychiatry. 2001 Sep;62(9):707-14. doi: 10.4088/jcp.v62n0908. PMID 11681767
- [Result] Yang YK, Nelson L, Kamaraju L, Wilson W, McEvoy JP. Nicotine decreases bradykinesia-rigidity in haloperidol-treated patients with schizophrenia. Neuropsychopharmacology. 2002 Oct;27(4):684-6. doi: 10.1016/S0893-133X(02)00325-1. PMID 12377405